CLINICAL TRIAL: NCT06170866
Title: Peer Partners to Improve Physical Activity in Older Latino and Latina Adults With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Cristina Colón-Semenza, Principal Investigator, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-117S-2; P30AG067988 (NIH)
Record Dates: First submitted 2023-11-10; First posted 2023-12-14 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Exercise; Peer Support; Hispanic; Parkinson´s Disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a prospective feasibility trial, single group pre-posttest design and it aims to enroll 20 participants. For this feasibility study, the sample size is comparable to other feasibility trials in populations of individuals with Parkinson disease (Lima & Rodrigues-de-Paula, 2013; Ellis et al., 2013, Colón-Semenza et al., 2018)17,19,20. This sample size will allow for a comparison in feasibility, acceptability, and appropriateness within and across groups. This sample will allow for identifying trends and preliminary efficacy for this intervention. This study will help to inform an appropriate sample size to adequately power larger samples in future studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social support for physical activity (Experimental): Socially supported (peer, family and group) physical activity group.
  Interventions: Behavioral: Socially supported physical activity

INTERVENTIONS:
Behavioral: Socially supported physical activity — Use of a culturally and linguistically tailored intervention that uses mobile health technology plus social support to increase engagement in physical activity in the management of Parkinson´s disease.

SUMMARY:
The goal of this interventional study is to culturally adapt and determine feasibility of the peer partner training program and the peer-supported mobile health physical activity intervention in older Latin/Hispanic people with Parkinson's disease.

The main question[s] it aims to answer are:

* What is the feasibility of the peer partner training program?
* What is the feasibility of the peer-supported mobile health physical activity intervention?
* What are the effects of the peer-supported mobile health physical activity intervention on physical activity, motivation, depression, apathy and self-efficacy?

Participants will be asked to:

* Wear a research-grade activity monitor, Actigraph GT9X device for 10 days at the beginning and end of the study.
* Watch 11 educational videos about Parkinson´s disease and exercise and attend two virtual educational sessions.
* Connect with another person with Parkinson´s disease one time a week on a virtual meeting platform for 8 weeks.
* Use Fitbit activity monitors and connect with other participants through the Fitbit application for 8 weeks.
* Attend a weekly online exercise class for 8 weeks with other people with Parkinon´s disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson disease,
* Able to walk without the assistance of another person for 10 minutes

  -≥ 29 on Telephone Interview for Cognitive Status (TICS)
* To have a close friend/family member over the age of 18 that would support the participant during the intervention

  -≥ 50 years of age
* Hispanic
* To be willing to use an activity monitor and use a Fitbit and Fitbit application
* To be on a stable course of PD medications without any plans for change over the next 3 months
* To be able to speak, read and write in Spanish or English

Exclusion Criteria:

* Unstable cardiopulmonary, orthopedic, psychological or metabolic condition
* Atypical Parkinsonism Disorders
* A fall in the last 6 months (that was unrelated to an external force)
* Currently engaging in 150 minutes of mod-vigorous physical activity/week

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Colón-Semenza, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng EM, Tonn S, Swain-Eng R, Factor SA, Weiner WJ, Bever CT Jr; American Academy of Neurology Parkinson Disease Measure Development Panel. Quality improvement in neurology: AAN Parkinson disease quality measures: report of the Quality Measurement and Reporting Subcommittee of the American Academy of Neurology. Neurology. 2010 Nov 30;75(22):2021-7. doi: 10.1212/WNL.0b013e3181ff96dd. PMID 21115958
- [Background] Rogers G, Davies D, Pink J, Cooper P. Parkinson's disease: summary of updated NICE guidance. BMJ. 2017 Jul 27;358:j1951. doi: 10.1136/bmj.j1951. No abstract available. PMID 28751362
- [Background] Alberts JL, Rosenfeldt AB. The Universal Prescription for Parkinson's Disease: Exercise. J Parkinsons Dis. 2020;10(s1):S21-S27. doi: 10.3233/JPD-202100. PMID 32925109
- [Background] Johansson ME, Cameron IGM, Van der Kolk NM, de Vries NM, Klimars E, Toni I, Bloem BR, Helmich RC. Aerobic Exercise Alters Brain Function and Structure in Parkinson's Disease: A Randomized Controlled Trial. Ann Neurol. 2022 Feb;91(2):203-216. doi: 10.1002/ana.26291. Epub 2022 Jan 19. PMID 34951063
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Marras C, Beck JC, Bower JH, Roberts E, Ritz B, Ross GW, Abbott RD, Savica R, Van Den Eeden SK, Willis AW, Tanner CM; Parkinson's Foundation P4 Group. Prevalence of Parkinson's disease across North America. NPJ Parkinsons Dis. 2018 Jul 10;4:21. doi: 10.1038/s41531-018-0058-0. eCollection 2018. PMID 30003140
- [Background] Van Den Eeden SK, Tanner CM, Bernstein AL, Fross RD, Leimpeter A, Bloch DA, Nelson LM. Incidence of Parkinson's disease: variation by age, gender, and race/ethnicity. Am J Epidemiol. 2003 Jun 1;157(11):1015-22. doi: 10.1093/aje/kwg068. PMID 12777365
- [Background] Damron L, Litvan I, Bayram E, Berk S, Siddiqi B, Shill H. Hispanic Perspectives on Parkinson's Disease Care and Research Participation. J Alzheimers Dis. 2021;81(2):809-819. doi: 10.3233/JAD-210231. PMID 33843687
- [Background] Fullard ME, Thibault DP, Hill A, Fox J, Bhatti DE, Burack MA, Dahodwala N, Haberfeld E, Kern DS, Klepitskava OS, Urrea-Mendoza E, Myers P, Nutt J, Rafferty MR, Schwalb JM, Shulman LM, Willis AW; Parkinson Study Group Healthcare Outcomes and Disparities Working Group. Utilization of rehabilitation therapy services in Parkinson disease in the United States. Neurology. 2017 Sep 12;89(11):1162-1169. doi: 10.1212/WNL.0000000000004355. Epub 2017 Aug 23. PMID 28835397
- [Background] Crespo CJ, Smit E, Andersen RE, Carter-Pokras O, Ainsworth BE. Race/ethnicity, social class and their relation to physical inactivity during leisure time: results from the Third National Health and Nutrition Examination Survey, 1988-1994. Am J Prev Med. 2000 Jan;18(1):46-53. doi: 10.1016/s0749-3797(99)00105-1. PMID 10808982
- [Background] Mantri S, Fullard M, Gray SL, Weintraub D, Hubbard RA, Hennessy S, Willis AW. Patterns of Dementia Treatment and Frank Prescribing Errors in Older Adults With Parkinson Disease. JAMA Neurol. 2019 Jan 1;76(1):41-49. doi: 10.1001/jamaneurol.2018.2820. PMID 30285047
- [Background] Hooker SP, Wilcox S, Rheaume CE, Burroughs EL, Friedman DB. Factors related to physical activity and recommended intervention strategies as told by midlife and older African American men. Ethn Dis. 2011 Summer;21(3):261-7. PMID 21942156
- [Background] Griffith DM, Bergner EM, Cornish EK, McQueen CM. Physical Activity Interventions With African American or Latino Men: A Systematic Review. Am J Mens Health. 2018 Jul;12(4):1102-1117. doi: 10.1177/1557988318763647. Epub 2018 Mar 20. PMID 29557237
- [Background] Callahan LF, Rivadeneira A, Altpeter M, Vilen L, Cleveland RJ, Sepulveda VE, Hackney B, Reuland DS, Rojas C. Evaluation of the Arthritis Foundation's Camine Con Gusto Program for Hispanic Adults With Arthritis. Hisp Health Care Int. 2016 Sep;14(3):132-40. doi: 10.1177/1540415316665202. Epub 2016 Aug 23. PMID 27553228
- [Background] Ige-Elegbede J, Pilkington P, Gray S, Powell J. Barriers and facilitators of physical activity among adults and older adults from Black and Minority Ethnic groups in the UK: A systematic review of qualitative studies. Prev Med Rep. 2019 Jul 13;15:100952. doi: 10.1016/j.pmedr.2019.100952. eCollection 2019 Sep. PMID 31367514
- [Background] Barcelona de Mendoza V, Damio G. Evaluation of a culturally appropriate peer coaching program for smoking cessation. Public Health Nurs. 2018 Nov;35(6):541-550. doi: 10.1111/phn.12542. Epub 2018 Sep 14. PMID 30596399
- [Background] Colon-Semenza C, Latham NK, Quintiliani LM, Ellis TD. Peer Coaching Through mHealth Targeting Physical Activity in People With Parkinson Disease: Feasibility Study. JMIR Mhealth Uhealth. 2018 Feb 15;6(2):e42. doi: 10.2196/mhealth.8074. PMID 29449201
- [Background] Dorsey ER, Constantinescu R, Thompson JP, Biglan KM, Holloway RG, Kieburtz K, Marshall FJ, Ravina BM, Schifitto G, Siderowf A, Tanner CM. Projected number of people with Parkinson disease in the most populous nations, 2005 through 2030. Neurology. 2007 Jan 30;68(5):384-6. doi: 10.1212/01.wnl.0000247740.47667.03. Epub 2006 Nov 2. PMID 17082464
- [Background] Lima LO, Rodrigues-de-Paula F. Recruitment rate, feasibility and safety of power training in individuals with Parkinson's disease: a proof-of-concept study. Braz J Phys Ther. 2013 Jan-Feb;17(1):49-56. doi: 10.1590/s1413-35552012005000069. English, Portuguese. PMID 23538458
- [Background] Ellis T, Latham NK, DeAngelis TR, Thomas CA, Saint-Hilaire M, Bickmore TW. Feasibility of a virtual exercise coach to promote walking in community-dwelling persons with Parkinson disease. Am J Phys Med Rehabil. 2013 Jun;92(6):472-81; quiz 482-5. doi: 10.1097/PHM.0b013e31828cd466. PMID 23552335
- [Background] Carvas Junior N, Gomes IC, Valassi JMR, Anunciacao L, Freitas-Dias R, Koike MK. Comparison of the printed and online administration of the Behavioral Regulation in Exercise Questionnaire (BREQ-2). Einstein (Sao Paulo). 2021 Aug 2;19:eAO6088. doi: 10.31744/einstein_journal/2021AO6088. eCollection 2021. PMID 34346988
- [Background] Bushnell DM, Martin ML. Quality of life and Parkinson's disease: translation and validation of the US Parkinson's Disease Questionnaire (PDQ-39). Qual Life Res. 1999 Jun;8(4):345-50. doi: 10.1023/a:1008979705027. PMID 10472167
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Mendoza-Vasconez AS, Marquez B, Benitez TJ, Marcus BH. Psychometrics of the self-efficacy for physical activity scale among a Latina women sample. BMC Public Health. 2018 Sep 5;18(1):1097. doi: 10.1186/s12889-018-5998-0. PMID 30185171
- [Background] Washburn RA, McAuley E, Katula J, Mihalko SL, Boileau RA. The physical activity scale for the elderly (PASE): evidence for validity. J Clin Epidemiol. 1999 Jul;52(7):643-51. doi: 10.1016/s0895-4356(99)00049-9. PMID 10391658
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Kadhim S, Pringsheim T, Le A, Fiest KM, Patten SB, Prisnie JC, Gill S, Bulloch AGM, Hu B, Jette N. Validating screening tools for depression in Parkinson's disease. Mov Disord. 2018 Jul;33(7):1184-1186. doi: 10.1002/mds.27371. Epub 2018 Mar 24. No abstract available. PMID 29573354
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Sockeel P, Dujardin K, Devos D, Deneve C, Destee A, Defebvre L. The Lille apathy rating scale (LARS), a new instrument for detecting and quantifying apathy: validation in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2006 May;77(5):579-84. doi: 10.1136/jnnp.2005.075929. PMID 16614016
- [Background] Leentjens AF, Dujardin K, Marsh L, Martinez-Martin P, Richard IH, Starkstein SE, Weintraub D, Sampaio C, Poewe W, Rascol O, Stebbins GT, Goetz CG. Apathy and anhedonia rating scales in Parkinson's disease: critique and recommendations. Mov Disord. 2008 Oct 30;23(14):2004-14. doi: 10.1002/mds.22229. PMID 18709683
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Noroozi A, Ghofranipour F, Heydarnia AR, Nabipour I, Shokravi FA. Validity and reliability of the social support scale for exercise behavior in diabetic women. Asia Pac J Public Health. 2011 Sep;23(5):730-41. doi: 10.1177/1010539509357342. Epub 2010 May 10. PMID 20460282

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Social support for physical activity
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Social Support for Physical Activity
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Disease duration [Mean (Standard Deviation); unit: years] | 8.2 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: A standardized measure of acceptability that indicates percent agreement with acceptability of the intervention ranging from 20-100%. Higher scores indicate agreement (better outcome) with the acceptability of the intervention.
Time Frame: After completion of the entire intervention (11 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | 93 (8.56)

2. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: A standardized measure of appropriateness that indicates percent agreement with appropriateness of the intervention ranging from 20-100%. Higher scores indicate more agreement (better outcome) with the appropriateness of the intervention.
Time Frame: After completion of the entire intervention (11 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | 89 (10.21)

3. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: A standardized measure of feasibility that indicates percent agreement with feasibility of the intervention ranging from 20-100%. Higher scores indicate more agreement (better outcome) with the feasibility of the intervention.
Time Frame: After completion of the entire intervention (11 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | 87 (11.11)

4. Secondary Outcome: Objective Measurement of Physical Activity
Description: Steps per day measured using a research-grade activity monitor will provide group mean change in physical activity from baseline to post-intervention.
Time Frame: 10 days at baseline and post-intervention (approximately 12 to 14 weeks)
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
steps/day | 110.77 (1891.27)

5. Secondary Outcome: Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2)
Description: The Behavioral Regulation in Exercise Questionnaire-2, Relative Autonomy Index, is a standardized, 19-item survey that evaluates motivation for exercise. The scores range from -24 to +20 with higher scores indicating increased motivation or better outcomes. The group mean change score is presented.
Time Frame: Baseline and post Intervention (approximately 12 to 14 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | 0.55 (1.96)

6. Secondary Outcome: Parkinson's Disease Questionnaire-39 (PDQ-39)
Description: The Parkinson's Disease Questionnaire-39 (PDQ-39) is a 39-item, self-report survey that assess quality of life. The scores range from 0-100 and a decrease indicates an improvement in quality of life. The group mean change total scores will be evaluated.
Time Frame: Pre and post intervention (approximately 12 to 14 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | -7.11 (8.98)

7. Secondary Outcome: Geriatric Depression Scale-Short Form
Description: The Geriatric Depression Scale (GDS) -15, is a 15-item self-report measure of depression in older adults. The score ranges from 0-15 with higher scores indicating higher levels of depression (worse outcome). Group mean change scores related to depression are reported.
Time Frame: Pre and post intervention (approximately 12 to 14 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social support for physical activity
Number analyzed (Participants) | 10
score on a scale | -1.15 (2.17)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: There was a systematic assessment of adverse event reporting by the research assistants that queried participants each week if they experienced an adverse event in the past week.
Arm/Group | Social support for physical activity
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT06170866/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT06170866/ICF_003.pdf